CLINICAL TRIAL: NCT06647485
Title: A Prospective Randomized Study for the Evaluation of the Impact of Point-by-Point Pulse Field Ablation on Autonomic Nervous System Modulation in Paroxysmal Atrial Fibrillation
Brief Title: Evaluation of the Impact of Pulsed Field Ablation on Autonomic Nervous System Modulation in Paroxysmal Atrial Fibrillation
Acronym: GPfIRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VZW Cardiovascular Research Center Aalst (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GPfIRE01-BWI-CS-012; CIV-24-02-046139-RS01 (Other: Eudamed)
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation (AF); Paroxysmal AF
Keywords: vagal modulation; ganglionated plexi; pulsed field; dual-energy focal ablation; paroxysmal atrial fibrillation; heart rate variability; pulmonary vein isolation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PF-only (Experimental): The PF-only arm includes patients with a clinical indication for ablation to manage their paroxysmal atrial fibrillation, who will undergo PVI using only PF energy
  Interventions: Procedure: PF-only PVI
- Hybrid (PF posterior/RF anterior) (Experimental): The Hybrid arm includes patients with a clinical indication for ablation to manage their paroxysmal atrial fibrillation, who will undergo PVI using both PF and RF energy
  Interventions: Procedure: Hybrid PVI
- RF-only (Active Comparator): The RF-only arm includes patients with a clinical indication for ablation to manage their paroxysmal atrial fibrillation, who will undergo PVI using only RF energy
  Interventions: Procedure: RF-only PVI

INTERVENTIONS:
Procedure: PF-only PVI — It consists in performing a point-by-point PVI using the Dual Energy THERMOCOOL SMARTTOUCH™ SF (DE STSF) ablation catheter with the TRUPULSE™ generator, employing only PF energy for ablation
  Arms: PF-only
Procedure: Hybrid PVI — It consists in performing a point-by-point PVI using the Dual Energy THERMOCOOL SMARTTOUCH™ SF (DE STSF) ablation catheter with the TRUPULSE™ generator, employing both PF and RF energy for ablation. Specifically, PF energy is used for the posterior segments and RF energy for the anterior segments of the pulmonary veins
  Arms: Hybrid (PF posterior/RF anterior)
Procedure: RF-only PVI — It consists in performing a point-by-point PVI using the Dual Energy THERMOCOOL SMARTTOUCH™ SF (DE STSF) ablation catheter with the TRUPULSE™ generator, employing only RF energy for ablation
  Arms: RF-only

SUMMARY:
The objective of this clinical trial is to evaluate the impact of pulse field (PF) energy, both alone and in combination with radiofrequency (RF) energy, on vagal modulation during point-by-point pulmonary vein isolation (PVI) in patients with paroxysmal atrial fibrillation (PAF). The effect of PF energy on ganglionated plexi (GP) will be assessed using heart rate variability (HRV) as a surrogate marker. Participants will be randomized into three groups: the PF-only group and the Hybrid group (PF posterior/RF anterior) as the experimental arms, and the RF-only group as the control arm. HRV will be measured before and 24 hours after the PVI procedure. Additionally, cardio and neuro biomarkers (Troponin and S100B) will be measured pre-procedure and 20 minutes post-ablation. All participants will be followed for 12 months, with 24-hour Holter-ECG evaluations scheduled at 3, 6, and 12 months after the initial ablation procedure.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic Paroxysmal Atrial Fibrillation (AF) that terminates spontaneously or with intervention within 7 days of onset
* Age range: 18-70 years
* Willing and capable of providing informed consent
* Able and willing to comply with all pre-, post-, and follow-up testing and requirements

Exclusion Criteria:

* Previously diagnosed Persistent AF (> 7 days in duration)
* Previous LA ablation
* Previous cardiac surgery
* Myocardial Infarction within the previous 3 months
* Severely compromised Left Ventricular Ejection Fraction (LVEF<40%)
* Presence of implanted pacemaker or Implantable Cardioverter-Defibrillator (ICD) or other implanted metal cardiac device that may interfere with the pulsed electric field energy
* Acute illness, active systemic infection, or sepsis
* Presence of intracardiac thrombus, myxoma, tumor, interatrial baffle or patch or other abnormality that precludes catheter introduction or manipulation.
* Severe mitral regurgitation
* Woman who are pregnant, lactating, or who are planning to become pregnant during the course of the clinical investigation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Acute HRV variation (PF-only vs. RF-only arm) | from enrolment to the day after the ablation procedure
  It is the acute difference in the HRV variation (Δ SDNN: baseline/1-day after ablation) between the PF-only arm and the control arm (RF-only).

SECONDARY OUTCOMES:
Acute HRV variation (Hybrid vs. RF-only arm) | from enrolment to the day after the ablation procedure
  The secondary endpoint is the acute difference in the HRV variation (Δ SDNN: baseline/1-day after ablation) between the Hybrid arm and the control arm (RF-only)

OTHER OUTCOMES:
Acute difference in biomarker release | Peri-procedural: from procedure start (after groin puncture) to its end (before sheaths removal)
  It measures the change in blood levels of the neuro-biomarker S100B (Δ S100B) and the cardiac injury biomarker Troponin (Δ Troponin), both measured before and immediately (~ 20 minutes) after the ablation
Atrial arrhythmia recurrences and atrial fibrillation burden | from day 91 to day 365 post-ablation
  It measures any difference between the study arms in terms of AT/AF/AFL documented recurrences and AF burden during the effective evaluation period (Day 91-Day 365)
Acute difference in resting Heart Rate (HR) | from enrolment to the day after the ablation procedure
  Acute difference in average resting HR (Δ HR: baseline/1-day after ablation) between the investigational arms compared to the control arm
HRV variation across the follow-up period | from the first follow-up (3-month) visit until the last one (12-month)
  It measures the HRV change at 3, 6 and 12 months after the ablation procedure to assess the durability of the vagal modulation

CONTACTS AND LOCATIONS:
Overall Officials: Tom De Potter, MD, Principal Investigator — Cardiovascular Research Center Aalst
Locations (1):
- OLV Hospital, Aalst, Belgium, Belgium

IPD SHARING:
Plan to Share IPD: No